CLINICAL TRIAL: NCT06971861
Title: Just ACT: School-Based Program Using Acceptance and Commitment Therapy (ACT) to Promote Student Well-being
Brief Title: Just ACT for Student Well-being
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: New Life Psychiatric Rehabilitation Association (Other)
Responsible Party: Principal Investigator, Amanda Kingsze CHEUNG, Research Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA240507
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Acceptance and Commitment Therapy; Psychological Well-being
MeSH Terms: conditions — Psychological Well-Being | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Group-based Acceptance and Commitment Therapy for youth delivered across four one-hour sessions
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The current program is based on ACT and consists of four one-hour sessions covering the six core components of psychological flexibility. The four sessions respectively focus on Cognitive Defusion, Being Present and Acceptance, Self-as-Context and Values, and Committed Action. All sessions involve experiential learning activities and reflective discussions. Each participant also receives a workbook to facilitate post-session home practice.
  Other Names: ACT

SUMMARY:
Most psychological conditions start developing during adolescent years. This makes adolescence an ideal and critical window for prevention efforts that help enhance stress management and mental health among the younger generations. This pilot study aims to develop a brief prevention program that focuses on youths' well-being and living as guided by their personal values.

ELIGIBILITY:
Inclusion Criteria:

* age of 35 years or below
* fluency in oral and written Chinese

Exclusion Criteria:

* active or current history of psychosis, bipolar disorder, or personality disorder
* active or current report of suicidal attempts
* active or current suicidal ideations for more than half the days
* any history of intellectual deficits

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2028-10-21 (Estimated); Study Completion 2028-10-21 (Estimated)

PRIMARY OUTCOMES:
Attendance | At the end of treatment
  Attendance across four sessions in percentage
Change in psychological flexibility as measured with the Multidimensional Psychological Flexibility Inventory | Before treatment, between the second and third session, within one week after treatment, and one month after treatment
  The Multidimensional Psychological Flexibility Inventory (MPFI; Rolffs et al., 2018) is the only validated measure that provides separate ratings on the six core processes of ACT (see Barrett et al., 2019). Items are rated on a 6-point Likert scale, from 1 - Never True to 6 - Always True, and averaged to obtain a score for each of the dimensions.

SECONDARY OUTCOMES:
Treatment retention | At the end of treatment
  Percentage of participants staying in treatment through the end
Change in well-being as measured with the Flourishing Scale | Before treatment, within a week after treatment, and one month after treatment
  The Flourishing Scale (FS) is an 8-item rating scale that measures sociopsychological prosperity, in terms of social relationships, purposeful or meaningful living, self-respect, and feeling of competence. Items are rated on a 7-point Likert scale, from 1 - Strong Disagreement to 7 - Strong Agreement.
Change in depressive symptoms as measured with Patient Health Questionnaire (PHQ-9) | Before treatment, within a week after treatment, and one month after treatment
  The nine-item Patient Health Questionnaire (PHQ-9; Kroenke & Spitzer, 2002) is a gold-standard measure of depressive symptoms an individual experienced in the prior two-week period. Items are rated on a 4-point Likert scale, from 0 - Not at All to 3 - Nearly Every Day. Total score on the PHQ-9 ranges from 0 to 27, with higher scores indicating more severe impact of depressive symptoms on an individual's life.
Change in anxiety symptoms as measured with the Generalized Anxiety Disorder (GAD-7) | Before treatment, within a week after treatment, and one month after treatment
  The seven-item Generalized Anxiety Disorder (GAD-7; Spitzer et al., 2006) is a gold-standard measure of anxiety symptoms an individual experienced in the prior two-week period. Items are rated on a 4-point Likert scale, from 0 - Not at All to 3 - Nearly Every Day. Total score on the GAD-7 ranges from 0 to 21, with higher scores indicating more severe impact of anxiety symptoms on an individual's life.
Treatment satisfaction | Within a week after treatment
  Participants are invited to rate on a 5-point Likert scale, from 1 - Strongly Disagree to 5 - Strongly Agree, designed specifically to assess their level of satisfaction with the intervention received in the current study. They are also asked in an open-ended way to provide qualitative feedback on the program, including their overall or any specific experience with the program not otherwise captured by the pre-set prompting questions.

CONTACTS AND LOCATIONS:
Locations (1):
- New Life Psychiatric Rehabilitation Association, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Sensitive data are collected and no authorization is obtained from participants